CLINICAL TRIAL: NCT01237717
Title: Relationship of Urine Sodium Excretion to Central Blood Pressure and Aortic Pulse Wave Velocity
Status: Completed | Type: Observational
Sponsor: DongGuk University (Other)
Collaborators: The Korean Society of Cardiology (Other)
Responsible Party: Principal Investigator, Moo-Yong Rhee, Professor, DongGuk University
Other Study IDs: 2010-1-15
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Hypertension
Keywords: hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, Plasma, and DNA sample (whole blood)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- normotensive subjects: subjects without hypertension, and without diabetes, ischemic heart disease, major arrhythmia, heart failure, secondary hypertension, high grade renal disease,
- Hypertensive subjects: subjects with hypertension,
  1. currently not treated at least within 6 months
  2. without diabetes, ischemic heart disease, major arrhythmia, heart failure, secondary hypertension, high grade renal disease,

SUMMARY:
One interesting area is the relationship of high salt intake and central aortic blood pressure. High salt intake is associated development of hypertension and cardiovascular mortality. Central aortic pressure is better correlated with cardiovascular events and mortality. With recent advances in technology, it is possible to measure central aortic pressure noninvasively and easily. Until now there is no study to evaluate the relationship of high salt intake and aortic blood pressure.

The purpose of the present study is to evaluate the relationship of high salt intake and aortic blood pressure and aortic stiffness.

Subjects with or without hypertension will be enrolled for investigation. Subjects with hypertension should be never treated with antihypertensive medications. Subjects with secondary hypertension, diabetes, heart failure, high grade kidney disease, ischemic heart disease, and major arrhythmia will be excluded.

Sodium intake is measured by 24 hour urinary sodium excretion, with the measurement of peripheral and central aortic blood pressure, and aortic pulse wave velocity.

Salt sensitive hypertension related single nucleotide polymorphism will be analyzed to define the relationship with high salt intake and aortic pressure and pulse wave velocity.

DETAILED DESCRIPTION:
Measurements: should be performed for 2 days

1. 24 hour urine Na, K and Creatinine, 24 hour urine amount

   1. Calculation of urine completeness index : Cr/(21 x Bwt)
   2. Definition of complete urine collection: complete index ≥ 0.7 and loss not more than one time and 100 mL
2. Peripheral blood pressure (pBP)

   1. Microlife WatchBP Office
   2. Sitting position
   3. After 5 minutes resting
   4. Peripheral systolic BP (pSBP), Peripheral diastolic BP (pDBP),
3. Central aortic blood pressure

   1. SphygmoCor (AtCor Medical, Australia)
   2. Central systolic blood pressure
   3. Difference between peripheral SBP and central SBP (SBPp-c)
4. Pulse wave velocity

   1. VP2000 (Colin, Japan)
   2. Central pulse wave velocity: carotid-femoral Pulse Wave Velocity
   3. Measure by tape
   4. distance from suprasternal notch to carotid artery
   5. distance from suprasternal notch to femoral artery
   6. Silent environment
5. Blood chemistry and complete blood count

   1. Measure at the morning of second day after overnight fasting
   2. complete blood count, blood urea nitrogen/Creatinine, fasting blood glucose, Total cholesterol, Triglyceride, High density lipoprotein cholesterol
6. 24 hour ambulatory blood pressure measurement

Measurement protocol

1. 1st day

   1. Visit hospital before 9:00 AM after overnight fasting
   2. start 24 hour urine collection from 9:00 AM (with education for complete collection)
   3. start 24 hour ambulatory blood pressure monitoring, in parallel with 24 hour urine collection
2. 2nd day

   1. Measure central aortic blood pressure
   2. Measure blood Lab
   3. Measure Pulse Wave Velocity

Analysis of Salt sensitive gene polymorphism

1. Single Base Extension technology(SBE)
2. single nucleotide polymorphism rs2398162 and other salt sensitive hypertension related single nucleotide polymorphism

ELIGIBILITY:
Inclusion Criteria:

* subjects without hypertension: n=100
* subjects with hypertension, not treated at least within 6months: n=100

Exclusion Criteria:

* secondary hypertension
* known diabetes (HbA1C >7.5%)
* night worker
* stage 3 hypertension
* renal artery stenosis
* primary aldosteronism
* elevated GOT and/or glutamate-pyruvate transaminase > 2 fold of normal range
* heart failure, significant arrhythmia, angina, myocardial infarction, stroke, carotid stenosis
* pregnancy
* autoimmune disease, debilitating disease
* significant liver disease; active hepatitis, liver cirrhosis
* alcoholics
* Renal disease: Cr > 1.2 and/or proteinuria
* Medication affecting blood pressure and/or vascular stiffness, including lipid lowering agents

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subjects with or without hypertension
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
the relationship between 24 hour ambulatory blood pressure and 24 hour urine sodium/potassium excretion | cross-sectional study
  the relationship between 24 hour ambulatory blood pressure and 24 hour urine sodium/potassium excretion will be analysed. daytime, nighttime and morning BP will be analysed to 24 hour urinary sodium/potassium excretion

SECONDARY OUTCOMES:
the relationship between 24 hour urinary sodium/potassium excretion and central BP and arterial stiffness | Cross-sectional study

OTHER OUTCOMES:
the relationship between ambulatory BP variability and arterial stiffness | Cross-sectional study

CONTACTS AND LOCATIONS:
Overall Officials: Moo-Yong Rhee, Prof,MD, PhD, Principal Investigator — Cardiovascular Center, Dongguk University Ilsan Hospital
Locations (1):
- Dongguk University Ilsan Hospital, Goyang, Gyenggi, South Korea